CLINICAL TRIAL: NCT01132222
Title: A Randomized, Open Label, 2-treatment, Single Dose, Crossover, Bioequivalence Study of Ibuprofen 200 mg+Pseudoephedrine HCL 30 mg Tablets of Dr. Reddy's and Advil® Cold and Sinus Caplets of Wyeth Consumer Healthcare Under Fed Conditions.
Brief Title: Bioequivalence Study of Ibuprofen 200 mg + Pseudoephedrine HCL 30 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: M.S. Mohan, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 431-04
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Ibuprofen and Pseudoephedrine
MeSH Terms: interventions — Ibuprofen; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen + Psuedoephedrine Hydrochloride (Experimental): Ibuprofen 200 mg + Pseudoephedrine HCL 30 mg Tablets
  Interventions: Drug: Ibuprofen + Pseudoephedrine Hydrochloride
- Advil® Cold and Sinus (Active Comparator): Advil® Cold and Sinus Tablets of Wyeth Consumer Healthcare
  Interventions: Drug: Ibuprofen + Pseudoephedrine Hydrochloride

INTERVENTIONS:
Drug: Ibuprofen + Pseudoephedrine Hydrochloride — Ibuprofen 200 mg + Pseudoephedrine Hydrochloride 30 mg Tablets
  Other Names: Advil® Cold and Sinus

SUMMARY:
The purpose of this study is to assess the bioequivalence of Ibuprofen 200 mg + Pseudoephedrine HCL 30 mg under fed conditions.

DETAILED DESCRIPTION:
This study assess the bioequivalence of Ibuprofen 200 mg + Pseudoephedrine HCL 30 mg Tablets of Dr. Reddy's and Advil® Cold and Sinus Caplets of Wyeth Consumer Healthcare in healthy human adult subjects with the single oral administration under fed conditions with a washout period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects between 18-50 years of age (inclusive), weighing as per the standard height and weight chart of Life Insurance Corporation of India (II Underweight and Overweight Min. & Max. Chart)
* Subjects who have no evidence of underlying disease during screening medical history and whose physical examination is performed within 21 days to commencement of the study.
* Subjects whose screening laboratory values are within normal limits or considered by the physician/Principal Investigator to be of no clinical significance.
* Informed consent given in written form according to section 10.3 of the protocol.
* Female Subjects:

  1. of child bearing potential practicing an acceptable method of birth control for the duration of study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
  2. postmenopausal for at least 1 year.
  3. surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject.

Exclusion Criteria:

1. History or presence of significant:

   i. Cardiovascular, pulmonary, hepatic, renal hematological; gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
   * Alcohol dependence, alcohol abuse or drug abuse within past one year.
   * Moderate to heavy smoking (> 10 cigarettes/day) or on assumption of tobacco products.
   * History of difficulty in swallowing.
   * Clinically significant illness within 4 weeks before the start of the study
   * Asthma, urticaria or other allergic type reactions after taking any medication.
2. Subjects who, through completion of the study, would have donated in excess of

   * 500 ml of blood in 14 days, or
   * 500 - 800 m l of blood in 14 days (unless approved by the Principal Investigator)
   * 1000 ml of blood in 90 days
   * 1250 ml of blood in 120 days
   * 1500 ml of blood in 180 days
   * 2000 ml of blood in 270 days
   * 2500 ml of blood in 1 year
3. Participation in another clinical trial within the preceding 28 days of study start.
4. Subjects who have:

   * Systolic blood pressure less than 90 mm of Hg and more than 150 mm of Hg
   * Diastolic blood pressure less than 60 m of Hg and more than 95 mm of Hg. Minor deviations (1-3 mm Hg) at check-in may be acceptable at the discretion of the physician/investigator
   * Pulse rate below 50/min. and above 105/min.
5. Female volunteers demonstrating a positive pregnancy screen or currently breast-feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2004-09; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Vijayanthi G, MBBS, MD, Principal Investigator — Lotus Labs Pvt. Ltd.
Locations (1):
- Lotus Labs Pvt. Ltd., Bangalore, Karnataka, India